CLINICAL TRIAL: NCT03854305
Title: Phase 2a Multicenter Randomized Double-Blind Placebo-Controlled Parallel Study to Evaluate the Efficacy and Safety of Oral PRV-6527 (JNJ-40346527), an Inhibitor of CSF-1 Receptor, in Subjects With Moderately to Severely Active Crohn's
Brief Title: Phase 2a Study of PRV-6527 in Subjects With Moderately to Severely Active Crohn's Disease
Acronym: PRINCE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Provention Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRV-6527-CD2a; 2017-003017-25 (EudraCT Number)
Record Dates: First submitted 2019-02-23; First posted 2019-02-26 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRV-6527 (Experimental): Oral administration, 2X daily for 12 weeks
  Interventions: Drug: PRV-6527
- Placebo (Placebo Comparator): Oral administration, 2X daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRV-6527 — Treatment
  Arms: PRV-6527
Drug: Placebo — Comparator
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of oral PRV-6527 in the treatment of moderately to severely active Crohn's disease

DETAILED DESCRIPTION:
This is a Phase 2a, randomized, double-blind, placebo-controlled, parallel-group, multicenter study in adult subjects with moderately to severely active Crohn's disease.

Eligible subjects include males and females aged 18-75 years with moderately to severely active CD for at least 3 months. Each subject will receive the assigned treatment over 12 weeks, followed by a 4-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be a man or woman between 18 years and 75 (inclusive) years of age.
2. Has moderate to severe CD and a histologic diagnosis of CD for at least 3 months before screening.

Exclusion Criteria:

1. Has other gastrointestinal inflammatory diseases.
2. Has any malignancy or lymphoproliferative disorder other than nonmelanoma cutaneous malignancies or cervical carcinoma in situ that has been treated with no evidence of recurrence.
3. Has colon cancer or severe dysplasia. Subjects with CD for ≥8 years involving the colon are not excluded if they had a colonoscopy to assess for the presence of dysplasia within 1 year before baseline or if they had a colonoscopy at the screening visit that excludes any evidence of malignancy.
4. Has current signs or symptoms of an acute infection or infected skin wounds or ulcers, with the exception of nonserious infections in the opinion of the Investigator (e.g. sepsis, pneumonia, or pyelonephritis), including any infection requiring hospitalization or IV antibiotics, within 8 weeks before baseline.
5. Has severe, progressive, or uncontrolled renal, hepatic, hematological, endocrine, pulmonary, cardiac, neurologic, cerebral, or psychiatric disease, or signs and symptoms thereof.
6. Has any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the subject (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline to Week 12 in Crohn's Disease Activity Index score | 12 weeks
  Crohn's Disease Activity Scale will be assessed by collecting information on 8 different Crohn's Disease-related variables : extra-intestinal manifestations, abdominal mass, weight, hematocrit, total number of liquid stood, abdominal pain/cramping, use of antidiarrheal drug(s) and/or opiates, and general well-being. The last 4 variable are based on dairy of patient for 7 days Scale range is 0 to 600 with 0 being the best oputcome and a score of 600, the worst outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Provention Bio, MD, Study Director — Provention Bio
Locations (51):
- Austria (5):
  - Clinical Site, Innsbruck
  - Clinical Site, Klagenfurt
  - Clinical Site, Sankt Pölten
  - Clinical Site, Sankt Veit an der Glan
  - Clinical Site, Vienna
- Germany (5):
  - Clinical Site, Berlin
  - Clinical Site, Hamburg
  - Clinical Site, Kiel
  - Clinical Site, Landshut
  - Clinical Site, Ulm
- Hungary (4):
  - Clinical Site2, Budapest
  - Clinical Site, Budapest
  - Clinical Site, Miskolc
  - Clinical Site, Mosonmagyaróvár
- Poland (8):
  - Clinical Site, Bydgoszcz
  - Clinical Site2, Krakow
  - Clinical Site, Krakow
  - Clinical Site, Lodz
  - Clinical Site, Piotrkow Trybunalski
  - Clinical Site, Warsaw
  - Clinical Site2, Wroclaw
  - Clinical site, Wroclaw
- Russia (10):
  - Clinical site, Kemerovo
  - Clinical Site, Krasnoyarsk
  - Clinical Site2, Moscow
  - Clinical Site, Moscow
  - Clinical Site, Penza
  - Clinical site, Rostov-on-Don
  - Clinical Site, Saint Petersburg
  - Clinical Site2, Samara
  - Clinical Site, Samara
  - Clinical Site, Tomsk
- Spain (4):
  - ClinicaL Site, Córdoba
  - Clinical Site, Girona
  - Clinical Site 2, Madrid
  - Clinical Site, Madrid
- Ukraine (15):
  - Clinical Site, Kharkiv
  - Clinical site, Khmelnytskyi
  - Clinical Site 3, Kyiv
  - Clinical Site2, Kyiv
  - Clinical Site, Kyiv
  - Clinical Site2, Lviv
  - Clinical Site, Lviv
  - Clinical Site, Odesa
  - Clinical Site, Ternopil
  - Clinical Site2, Vinnytsia
  - Clinical Site3, Vinnytsia
  - Clinical Site, Vinnytsia
  - Clinical Site2, Zaporizhzhya
  - Clinical Site3, Zaporizhzhya
  - Clinical Site, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No